CLINICAL TRIAL: NCT01379716
Title: Immunolabeling Evaluation of Five Selected Markers in Skin Biopsies of Patients With Postherpetic Neuralgia (PHN) and Age and Gender-Matched Normal Controls
Brief Title: Evaluation of Five Selected Markers in Skin Biopsies of Patients With Postherpetic Neuralgia and Healthy Controls
Acronym: STTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Charles Argoff, Principal Investigator, Albany Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INT/AMC-001
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Postherpetic Neuralgia; Healthy Age/Gender Matched Volunteers
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: skin biopsy — Using a punch biopsy, the study doctor will take a small sample of skin (3mm diameter) from a pre-defined site of the subject. For PHN patients, 4 biopsies will be obtained: 2 in an area of PHN and 2 in a contralateral control site. Biopsy sites for each PHN control subject will be matched anatomically to the corresponding PHN patient with two biopsies each from symmetrical sites in a left and right dermatome. One biopsy from each site in each subject will be fixed in a left and right dermatome. One biopsy from each site in each subject will fixed yb immersion in 4% paraformaldehyde for immunocytochemical analysis, and the second biopsy form each site will be flash frozen for assessments of mRNA expression.

SUMMARY:
Postherpetic Neuralgia is a painful nerve condition that can occur when nerve fibers are damaged following an outbreak of shingles.

The purpose of this study is to identify and study abnormalities in the nerves and cells in the of patients with postherpetic Neuralgia (PHN) and characterize changes that could be responsible for causing nerve pain. This data will be compared to the tissue of healthy volunteers. Our goal is that this information will lead to the development of better treatment options for people with painful nerve conditions.

ELIGIBILITY:
Inclusion Criteria:

Group 1: 5 Caucasian males >50 years of age with PHN of greater than 6 months duration since rash healed and clinically meaningful pain (Visual Analog Scale (VAS) >40mm at Baseline) Group 2: 5 Caucasian males >50 years of age, non-diabetic with no nervous system disease (healthy control groups)

Exclusion Criteria:

1. History of clinically significant liver disease, serious peripheral vascular disease, a blood clotting disorder, or any other medical condition felt to be exclusionary by the investigator
2. Allergy to lidocaine
3. Unwillingness to sign informed consent or any other reasons for which the investigator feels the subject cannot complete the study
4. History of slow-healing diabetic foot ulcers
5. HgA1c >11% within the last three months
6. Active cancer within the previous two years, except treated basal cell carcinoma of the skin
7. Co-morbidities that can produce neuropathy
8. Subjects taking sodium channel blockers within one week of study treatment and throughout the study
9. Subjects taking any other experimental drugs within 30 days prior to enrollment
10. Application of lidocaine patch to either foot or to PHN site within two weeks of enrollment

Ages: 50 Years to 95 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
use of genetic data to enhance the search for targeted therapeutic approaches to chronic pain management | One year
  The skin biopsies will be used to identify the site of expression of selected makers in skin, including nerve fibers and skin substructures in patients with PHN and age and gender-atched normal controls.

CONTACTS AND LOCATIONS:
Overall Officials: James P. Wymer, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States